CLINICAL TRIAL: NCT05906537
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of SKB410 for Injection in Subjects With Advanced Solid Tumors
Brief Title: SKB410 for Injection in Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan Kelun Pharmaceutical Research Institute Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SKB410-I-01
Record Dates: First submitted 2023-05-16; First posted 2023-06-18 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dose Escalation (Experimental): Several dose levels are planned in the study and administered every 2 weeks.
  Interventions: Drug: SKB410 for injection

INTERVENTIONS:
Drug: SKB410 for injection — SKB410 for injection is administered every 2 weeks (q2w) until radiographic disease progression (PD), intolerable toxicity, death, or discontinuation of treatment, whichever occurs first.

SUMMARY:
This is a multicenter, open-label, multiple-dose dose finding and expansion study to evaluate the safety, tolerability, pharmacokinetic(PK) profile, and anti-tumor efficacy of SKB410 for injection in patients with advanced solid tumors.

DETAILED DESCRIPTION:
This is a multicenter, open-label, multiple-dose dose finding and expansion study to evaluate the safety, tolerability, PK profile, and anti-tumor efficacy of SKB410 for injection in patients with advanced solid tumors.This is a dose escalation study , and subjects with advanced solid tumors will be enrolled to receive SKB410 for Injection.

ELIGIBILITY:
Inclusion Criteria:

1. At the time of signing the ICF: age ≥ 18 years, male or female.
2. Subjects with histologically or cytologically confirmed locally advanced or metastatic solid tumors who have failed/are intolerant/ineligible to or do not have standard therapy, and have at least one measurable lesion meeting Response Evaluation Criteria in Solid Tumors (RECIST v1.1).
3. Eastern Cooperative Oncology Group (ECOG) score of 0 to 1.
4. Expected survival ≥ 3 months.
5. Subjects with adequate organ and bone marrow function confirmed by laboratory results within 3 days prior to the first dose.
6. Subjects of childbearing potential (male or female) must use effective medical contraception during the study and continue contraception until 210 days after the last dose for female subjects and until 120 days after the last dose for male subjects.
7. Ability to understand and willingness to sign ICF, and will be able to comply with the protocol-specified visits and relevant procedures.

Exclusion Criteria:

1. Has received anti-tumor therapy, including chemotherapy, targeted therapy, tumor immunotherapy, and traditional Chinese medicinal products with anti-tumor indications, within 4 weeks prior to the first dose or within 5 half-lives of known drugs (whichever is shorter).
2. Has received radiotherapy within 4 weeks prior to the first dose.
3. Has had major surgery within 4 weeks prior to the first dose.
4. Has received strong cytochrome P450 (CYP3A4) inhibitors or inducers (see Annex 4) within 2 weeks prior to the first dose or within 5 half-lives of known drug, whichever is longer.
5. Has not recovered to normal or ≤ Grade 1 from any AE and/or complication due to any prior therapy (except alopecia or pigmentation).
6. Has known history of allergy to any component of SKB410 or other monoclonal antibodies.
7. Has a known previous or concurrent other malignancies within 5 years prior to signing the ICF.
8. Presence of active central nervous system (CNS) metastases and/or carcinomatous meningitis.
9. Has active autoimmune disease with systemic therapy or immunosuppressive therapy within 2 years prior to signing the ICF.
10. Has uncontrolled or severe cardiovascular disease.
11. Has uncontrolled systemic diseases.
12. Presence of clear neurological or psychiatric disorder.
13. Has active infection requiring systemic.
14. Has human immunodeficiency virus (HIV) infection; has any active viral hepatitis.
15. Pregnant or lactating.
16. Has prior autologous/allogeneic hematopoietic stem cell transplantation or solid organ transplantation.
17. Has any other conditions such as medical history, treatment and laboratory abnormalities that may confound the study results, interfere with the subject's compliance, or impair the subject's interests, as assessed by the investigator or the sponsor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-06-30 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of subjects achieving Dose-limiting toxicity (DLT) | From data of initial dose until up to 28 days for treatment
  DLT is defined as an adverse event (AE) that meets protocol defined DLT criteria during cycle 1 and is at least possibly related to study drug.
Maximum Tolerated Dose (MTD) | From data of initial dose until up to 28 days for treatment
  MTD refers to the highest dose at which the subject's DLT incidence meets the EWOC principle (probability of DLT incidence exceeding 33% is less than 25%) during the DLT observation period.

OTHER OUTCOMES:
ORR | through study completion, an average of 2 years
  ORR: it refers to the proportion of subjects with best response of CR or PR after treatment.
DCR | through study completion, an average of 2 years
  DCR: it refers to the proportion of subjects with best response of response (PR + CR) and SD after treatment.
DOR | through study completion, an average of 2 years
  DOR: it refers to the time from the subject's first assessment of CR or PR to disease progression or death due to any cause.
PFS | through study completion, an average of 2 years
  PFS: it refers to the time from the start of treatment until disease progression (PD) or death.
OS | through study completion, an average of 2 years
  OS: it refers to the time from the first dose to death due to any cause (the last follow-up time for subjects who are lost to follow-up; the end of follow-up date for subjects who are still alive at the end of the study).

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No